CLINICAL TRIAL: NCT00345982
Title: Augmenting Clozapine With Sertindole - a Double Blinded Randomized Placebo Study
Brief Title: Augmenting Clozapine With Sertindole - SERCLOZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Jimmi Nielsen, M.D, Aalborg Psychiatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2005/150
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Last update posted 2010-09-27 (Estimated); Status verified 2010-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Treatment-resistant; sertindole; clozapine
MeSH Terms: conditions — Schizophrenia | interventions — sertindole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Sertindole 16 mg
  Interventions: Drug: Serdolect
- B (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Serdolect — 16 mg, 12 weeks
  Other Names: sertindole
  Arms: A
Drug: placebo — placebo
  Arms: B

SUMMARY:
The purpose of the study is to determine whether addition of sertindole to clozapine treatment can improve psychosis or the metabolic side-effects of clozapine in patients with treatment-resistant schizophrenia.

DETAILED DESCRIPTION:
Around 20 % of patients with schizophrenia are treatment-resistant. Clozapine is still the drug of choice for these patients but 2/3 will not respond adequately to clozapine. In the study clozapine treatment is augmented with sertindole. Patients are randomized to either clozapine or sertindole for 12 weeks and continue in a open-label study with sertindole for 12 weeks. The purpose of the open-label study is to determine whether clozapine dosage can be reduced due to the addition of sertindole.

ELIGIBILITY:
Inclusion Criteria:

* ICD10 diagnosis of schizophrenia (F20.0-3)
* Clozapine treatment minimum 6 months
* Total PANSS >65
* No antipsychotic other than clozapine drug 1 month prior inclusion

Exclusion Criteria:

* QTc >500 ms
* Violence to SPC of clozapine or Serdolect
* Major depression
* Significant substance misuse interfering with participating in the study
* Cardiovascular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
PANSS total score | 12 weeks

SECONDARY OUTCOMES:
GAF | 12 weeks
WHOQOL-BREF | 12 weeks
CGI | 12 weeks
DAI | 12 weeks
Cognitive test | 12 weeks
Fasting glucose | 12 weeks
Lipids | 12 weeks
Hb1Ac | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jimmi Nielsen, M.D., Principal Investigator — Aalborg Psychiatric Hospital
Locations (1):
- Aalborg Psychiatric Hospital, Aalborg, Denmark

REFERENCES:
- [Derived] Nielsen J, Emborg C, Gydesen S, Dybbro J, Aagaard J, Haderup K, Glyngdal P, Fabricius S, Thode D, Lublin H, Andersen T, Damkier P, Taylor D. Augmenting clozapine with sertindole: a double-blind, randomized, placebo-controlled study. J Clin Psychopharmacol. 2012 Apr;32(2):173-8. doi: 10.1097/JCP.0b013e318248dfb8. PMID 22367659
- [Derived] Nielsen RE, Levander S, Thode D, Nielsen J. Effects of sertindole on cognition in clozapine-treated schizophrenia patients. Acta Psychiatr Scand. 2012 Jul;126(1):31-9. doi: 10.1111/j.1600-0447.2012.01840.x. Epub 2012 Feb 22. PMID 22356584